CLINICAL TRIAL: NCT03486652
Title: Rheumatological Manifestations in Inflammatory Bowel Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mustafa badary, Principal investigator, Assiut University
Other Study IDs: IBD
Record Dates: First submitted 2018-01-23; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IBD-related arthropathy is one of a group of inflammatory arthritides considered as seronegative spondyloarthropathies, a group of disorders that also includes ankylosing spondylitis, psoriatic arthritis, reactive arthritis, and undifferentiated SpA. IBD-related SpA is mainly characterized by axial involvement but may also be associated with peripheral symptoms, such as synovitis, dactylitis, or enthesitis

ELIGIBILITY:
Inclusion Criteria:

* any patient with inflammatory bowel diseases complaining of rheumatological manifestations

Exclusion Criteria:

* chronic hepatitis (c) patients
* Rheumatoid factor positive patients
* psoriatic patients.
* systemic lupus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with inflammatory bowel diseases complaining of rheumatological manifestations clinical examination with espicial emphysis on the joints.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
the prevalence of rheumatological manifestations in cases of corhn's and ulcerative colitis | one year
  evaluation of all cases for manifestations of rheumatological manifestations